CLINICAL TRIAL: NCT04019418
Title: Carbohydrate Intake and Gut Hormone Release During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18HH4889
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: carbohydrate; exercise; PYY; GLP-1; ghrelin; hormones
MeSH Terms: conditions — Obesity; Motor Activity | interventions — maltodextrin; Carbohydrates; Exercise; RE1-silencing transcription factor; Water

STUDY DESIGN:
Intervention Model Description: Participants perform all four trials in a randomized order
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be masked to the contents of the beverage. They will not be masked to whether it is a resting or exercise condition as this is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Carbohydrate Drink + Rest (Placebo Comparator): Participants will consume the no carbohydrate drink (300ml water) followed by a rest session
  Interventions: Other: Rest; Other: Water
- No Carbohydrate Drink + Exercise (Active Comparator): Participants will consume the no carbohydrate drink (300ml water) followed by an exercise session (75% VO2 max on a cycle ergometer)
  Interventions: Other: Exercise; Other: Water
- Carbohydrate Drink + Rest (Active Comparator): Participants will consume the carbohydrate drink (300ml water + 75g maltodextrin) followed by a rest session
  Interventions: Dietary Supplement: Maltodextrin (carbohydrate); Other: Rest
- Carbohydrate Drink + Exercise (Experimental): Participants will consume the carbohydrate drink (300ml water + 75g maltodextrin) followed by an exercise session (75% VO2 max on a cycle ergometer)
  Interventions: Dietary Supplement: Maltodextrin (carbohydrate); Other: Exercise

INTERVENTIONS:
Dietary Supplement: Maltodextrin (carbohydrate) — A drink containing 300ml of water and 75g of maltodextrin
  Arms: Carbohydrate Drink + Exercise; Carbohydrate Drink + Rest
Other: Exercise — 30 minutes on a cycle ergometer working at 75% VO2 max
  Arms: Carbohydrate Drink + Exercise; No Carbohydrate Drink + Exercise
Other: Rest — 30 minutes laying on a bed
  Arms: Carbohydrate Drink + Rest; No Carbohydrate Drink + Rest
Other: Water — A drink containing 300ml of water
  Arms: No Carbohydrate Drink + Exercise; No Carbohydrate Drink + Rest

SUMMARY:
It is well known that following a single session of moderate-to-high intensity exercise individuals experience a temporary suppression of hunger and a delay in the commencement of eating. This effect is believed to be due to changes in blood concentrations of specific hormones released from the gut that influence appetite.

Individuals undertaking physical activity often consume foods immediately before exercise in order to improve their performance. However, it is currently unknown whether this eating practice influences the gut hormone response to exercise as well as how hungry an individual feels post-exercise.

Therefore, the aim of this study is to investigate the effect of consuming a sugary (carbohydrate) drink immediately before starting an exercise session on the concentration of these gut hormones as well as the amount of food eaten in the hours following exercise completion.

DETAILED DESCRIPTION:
It is well established that following an acute bout of moderate-to-high intensity exercise individuals experience a transient suppression of hunger and a delay in the commencement of eating - a phenomenon referred to as exercise-induced anorexia. Acute exercise modulates the concentrations of gut hormones known to influence satiety, including the anorexigenic hormones glucagon-like peptide 1 (GLP-1) and peptide tyrosine tyrosine (PYY), as well as the acylated form of the orexigenic hormone ghrelin. These alterations in gut hormone concentrations have consequently been hypothesised to play a key role in exercise-induced anorexia.

Despite suppressing hunger and delaying eating, acute exercise does not appear to alter short-term energy intake in the immediate hours following exercise completion. The absence of a compensatory response therefore creates an energy deficit capable of inducing weight loss. Strategies that augment the gut hormone response to acute exercise may thus increase the potency of exercise as a weight-loss tool.

Research investigating the effect of exercise on appetite has frequently utilised participants in a fasting state. Undertaking exercise in this physiological condition contradicts current practices, as athletes often consume a carbohydrate source immediately prior to exercise in an attempt to maximise performance. It is currently unknown as to whether the consumption of carbohydrate during this period may further enhance the gut hormone response to exercise, and thus research into a potential additive effect is warranted.

High-intensity exercise increases sympathetic nervous system activity and catecholamine release. Catecholamine concentrations are negatively correlated with acylated ghrelin concentrations and may directly stimulate GLP-1 and PYY release via activation of β-receptors located on L-cells. The decrease in gastric emptying rate that is observed during high-intensity exercise is also attributed to this increase in sympathetic activity. Consequently, an increase in sympathetic nervous system activity has been postulated as a key mechanism underlying exercise-induced changes in gut hormone concentrations. However, to our knowledge, no study has directly measured the relationship between sympathetic nervous system activity and anorexigenic gut hormone release during exercise.

Therefore, the aim of this study is to examine any potential additive effects of carbohydrate ingestion immediately prior to exercise on gut hormone release and post-exercise appetite suppression. Furthermore, this study will look to investigate the mechanisms underlying changes in gut hormone concentrations experienced during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18-40 years (inclusive)
* Body mass index (BMI) of 18-30 kg/m2
* Willingness and ability to give written informed consent and willingness and ability to understand, to participate and to comply with the study requirements

Exclusion Criteria:

* Abnormal ECG
* Screening blood results outside of normal reference values
* Current smokers
* Current or history of substance abuse and/or excess alcohol intake
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* Started new medication within the last 3 months likely to interfere with energy metabolism, appetite regulation and hormonal balance, including: anti-inflammatory drugs or steroids, antibiotics, androgens, phenytoin, erythromycin or thyroid hormones.
* Participation in a research study in the 12 week period prior to entering this study.
* Any blood donation within the 12 week period prior to entering this study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 12 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Changes in GLP-1 concentration | During the study visit, 165 minutes
  Changes in GLP-1 concentration between exercise and resting conditions, and between carbohydrate and control conditions
Changes in PYY concentration | During the study visit, 165 minutes
  Changes in PYY concentration between exercise and resting conditions, and between carbohydrate and control conditions
Changes in acylated ghrelin concentration | During the study visit, 165 minutes
  Changes in acylated ghrelin concentration between exercise and resting conditions, and between carbohydrate and control conditions

SECONDARY OUTCOMES:
Changes in energy intake | During the study visit, 165 minutes
  Differences in energy intake at an ad libitum meal between exercise and resting conditions, and between carbohydrate and control conditions
Changes in Energy expenditure | During the study visit, 165 minutes
  Differences in energy expenditure between exercise and resting conditions, and between carbohydrate and control conditions.
Changes in energy balance | During the study visit, 165 minutes
  Differences in energy balance between exercise and resting conditions, and between carbohydrate and control conditions.
Glucose homeostasis | During the study visit, 165 minutes
  Changes in glucose homeostasis between exercise and resting conditions, and between carbohydrate and control conditions.
Changes in subjective nausea | During the study visit, 165 minutes
  Changes in subjective feelings of nausea as measured by visual analogue scales between exercise and resting conditions, and between carbohydrate and control conditions. Visual analogue scales will range from 0 mm to 100 mm with a higher score indicating a higher degree of nausea.
Changes in subjective appetite | During the study visit, 165 minutes
  Changes in subjective feelings of appetite as measured by visual analogue scales between exercise and resting conditions, and between carbohydrate and control conditions. Visual analogue scales will range from 0 mm to 100 mm with a higher score indicating a higher degree of fullness.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chambers, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available

REFERENCES:
- [Result] Frampton J, Serrano-Contreras JI, Garcia-Perez I, Franco-Becker G, Penhaligan J, Tan ASY, de Oliveira ACC, Milner AJ, Murphy KG, Frost G, Chambers ES. The metabolic interplay between dietary carbohydrate and exercise and its role in acute appetite regulation in males: a randomized controlled study. J Physiol. 2023 Aug;601(16):3461-3480. doi: 10.1113/JP284294. Epub 2023 Jun 15. PMID 37269207